CLINICAL TRIAL: NCT06214884
Title: Study Protocol: A Randomized Controlled Trial of a Mindfulness Intervention to Reduce Low Back Pain, Psychological Symptoms and Enhance Work Productivity Among Academic Staff in Malaysian Tertiary Education
Brief Title: Mindfulness Intervention to Reduce Low Back Pain Among Academicians
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Eva Zamri, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 304/CIPPT/6315622
Record Dates: First submitted 2023-12-26; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Low Back Pain
Keywords: mindfulness; low back pain; work productivity; anxiety; depression
MeSH Terms: conditions — Low Back Pain; Anxiety Disorders; Depression | interventions — Mindfulness; Proto-Oncogene Proteins c-raf

STUDY DESIGN:
Intervention Model Description: A single blind, parallel cluster randomized controlled trial will be conducted on 86 academic staff working in the tertiary education in Northern Region, West Coast of Peninsular Malaysia. At baseline, all participants must undergo the screening criteria for inclusion which are academic staff with moderate to severe symptom of anxiety with cut-off score of 16, mild to severe symptoms of depression with cut-off score of 16, and pain intensity of LBP should be at least >35mm using Visual analogue scale (VAS). Participants will be randomized at cluster level to receive either mindfulness intervention or control group. The intervention will be given for 5 sessions weekly for 60 minute/session. Outcome measures such as LBP, depression and anxiety symptoms, and work productivity will be measured at baseline and after 5-weeks. The control group will be given delayed treatment for 2 weeks after the trial ended.
Who Masked: Participant
Masking Description: Eligible participants were invited to participate in the interventional study. Their participation must be voluntarily. Those who agreed to participate will be randomized either to the intervention and wait-list control group. The participants will remain unaware of their group assignment, as the randomization sequence will be generated using computer-based randomization. This is known as single-blind study. Allocation will follow a 1:1 ratio, overseen by a researcher with no other involvement in this trial. The participants' names will be matched with the random number sequence. Clusters of participants were in the same workplace to avoid contamination of the intervention and enhance compliance within the intervention group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness for All (MFA) Group (Experimental): This intervention program named "MINDFULNESS FOR ALL (MFA)" developed on the conceptual basis of traditional mindfulness programs. Its formal structure resembles the traditional mindfulness programs, but it has been tailored to meet the needs and demands of employees.The MFA will take place in a group setting with 10-15 participants per cluster. Due to participants' convenience, the delivery mode of each intervention session would be conducted online. At the end of session, they will be provided the task and supplementary materials (e-book, short audio, and video) to be apply after the session.
  The modules will be delivered by two trainees. Both trainees have received the certificates from the mindfulness-based strategic awareness training course. Participants in the intervention group will be joining the modules for 5 sessions weekly for 60-minute/session. Details on the modules can be referred in the Supplement material.
  Interventions: Behavioral: Mindfulness for All
- Wait-list control group (Active Comparator): The wait-list control group will receive their training two weeks after interventional group complete their training. There will be a 90-minute online training session aimed at introducing participants to mindfulness in general and encouraging them to practice mindfulness by teaching several techniques. There will be no potential harm occurs among the subjects in the wait-list control group.
  Interventions: Behavioral: Mindfulness for All

INTERVENTIONS:
Behavioral: Mindfulness for All — Experimental:
  The MFA will take place in a group setting with 10-15 participants per cluster. Due to participants' convenience, the delivery mode of each intervention session would be conducted online. At the end of session, they will be provided the task and supplementary materials (e-book, short audio, and video) to be apply after the session. The modules will be delivered by two trainees. Both trainees have received the certificates from the mindfulness-based strategic awareness training course. Participants in the intervention group will be joining the modules for 5 sessions weekly for 60-minute/session. Details on the modules can be referred in the Supplement material.

SUMMARY:
Mindfulness interventions are a well-known approach for improving mental health. Nevertheless, the available evidence regarding their efficacy in addressing musculoskeletal pain (MSP) is limited, despite numerous studies demonstrating an association between psychological factors and MSP. Both mental health issues and MSP are prevalent among academicians, yet there is a scarce study on the application of mindfulness interventions to these specific concerns. Therefore, this study aimed to provide a study protocol that will focus on assessing the impact of mindfulness interventions on alleviating low back pain (LBP) symptoms, psychological symptoms, and improving work productivity among academic staff.

DETAILED DESCRIPTION:
This study acknowledges the significance of mindfulness interventions, primarily introduced by Jon Kabat-Zinn. Mindfulness, rooted in various religious traditions, has been associated with improved well-being. The efficacy of mindfulness interventions in addressing anxiety and mood disorders is supported by meta-analyses, indicating moderate effectiveness. The focus then shifts to workplace interventions, noting a rising trend in research on mindfulness from 2012 to 2022. Studies highlight its efficacy not only in mental health aspects among employees but also in reducing musculoskeletal disorders.

Previous studies revealing the positive impact of mindfulness on chronic musculoskeletal pain, psychological well-being, and overall health-related quality of life among nurses. Another study in Denmark combines mindfulness with physical and cognitive elements, demonstrating reductions in pain intensity across various body regions. While mindfulness in the workplace is well-explored, its application in academia, particularly among university teachers, is relatively new. Previous scoping review explores various psychological interventions, including Mindfulness-Based Interventions, cognitive behavioural therapy (CBT), and yoga, to reduce stress and burnout among teachers, but cautions against generalizing these findings to academicians due to the heterogeneity of their work nature.

Based on the fact mentioned above, it is imperative to initiate mindfulness interventions among the academicians targeting to reduce low back pain, psychological symptoms and enhance work productivity. As of our latest information, there are no existing programs accessible for this specific implementation in Malaysia. The specific objectives for this trial were as follows

1. To identify the efficacy of the mindfulness intervention in reducing the pain intensity of LBP among academic staffs.
2. To identify the efficacy of the mindfulness intervention in reducing depression and anxiety symptoms among academic staffs.
3. To identify the efficacy of the mindfulness intervention in improving work productivity among academic staffs.

ELIGIBILITY:
Inclusion criteria

* All academic staff aged 28-50 years old
* Able to understand Malay language
* Reported moderate to severe symptom of anxiety with cut-off score of 16,
* Reported mild to severe symptoms of depression with cut-off score of 16
* Presence of LBP during past month with pain intensity should be at least >35mm using Visual analogue scale (VAS).

Exclusion Criteria:

* Pregnancy or had planned to become pregnant in the coming months,
* History of trauma or accidents in the spinal region
* Medically diagnosed with congenital anomaly of the spine, rheumatoid arthritis, infections of the spine or discs, ankylosing spondylitis, spondylolisthesis, spondylosis, spinal tumor, systemic lupus erythymatosus, or osteoporosis.
* Had performed either spinal, intra-abdominal or femoral surgery.

Ages: 28 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Low back pain occurrence | Pre (week 0), Post intervention (week 5) and Follow-up (week 18)
  The questions about musculoskeletal pain focused on seven anatomical sites will be adapted based on the Nordic Musculoskeletal Questionnaire. The seven anatomical sites include low back, neck, right or/and left shoulder, right or/and left elbow, right or/and left wrist/hand and right or left knee, and right or left ankle with the binary response (yes/no). The instrument has an acceptable psychometric property and widely applied in Malaysian working population.
  During the screening process, participants will be asked whether they had experienced on low back pain during the past months that had lasted for longer than a day which were illustrated diagrammatically.
  After the intervention, the occurrence of low back pain pain will be re-assessed by asking whether they had experienced pain for each anatomical site, during the past months that had lasted for longer than a day which were illustrated diagrammatically.
Low back pain intensity | Pre (week 0), Post intervention (week 5) and Follow-up (week 18)
  Visual Analogue Scale (VAS) will be used to measure the participants' pain intensity during the pre and post-test. A VAS is commonly presented with unidimensional line, usually 100-mm long, starts from 0 'no pain' to 100 'severe intolerable pain'. Participants who reported pain at each anatomical site will be further asked to indicate which point along the line best represents their pain intensity.

SECONDARY OUTCOMES:
Psychological symptoms (anxiety) | Pre (week 0), Post intervention (week 5) and Follow-up (week 18)
  A Malay translated version of Beck Anxiety Inventory (BAI) consists of 21 items will be utilized in this study to assess the anxiety symptoms. The participants need to respond each item on a four-point Likert scale, ranging from 0 "not at all" to 3 "severely". The range of total scores is from 0 to 63, with higher numbers suggesting greater degrees of anxiety. The recommended clinical classification of scoring results are as follows: 0-7 suggests minimal anxiety, 8-15 suggests mild anxiety, 16-25 suggests moderate anxiety, and 26-63 suggests severe anxiety. According to the manual, the suggested cut-off for clinically significant anxiety on the BAI is 16. Previous local study has shown that the BAI-Malay version has excellent internal consistency (α=.92) and high test-retest reliability (r=.75).
Psychological symptoms (depression) | Pre (week 0), Post intervention (week 5) and Follow-up (week 18)
  A Malay translated version of Beck Depression Inventory (BDI) will be used to assess the depression symptoms. It consists of 21 items and for each item need to answer on a four-point Likert scale, ranging from 0 to 3. Each item were asked about the unique symptoms of depression which more reflective of the diagnostic criteria that are described by the American Psychiatric Association (APA). The possible range of total score is between 0 - 63. Then, the total score can be categorized into three group which reflect the severity levels: 0-10 points for "not depressed", 11-17 points for "mild to moderately depressed", and 18-63 points for "clinically relevant depression". Previous study indicated that the current Malay version of the BDI-II is psychometrically strong and appropriate for use in assessing depressive symptomatology among Malaysian.
Absenteeism and Presenteeism | Pre (week 0), Post intervention (week 5) and Follow-up (week 18)
  This study adapted an instrument known as Work Productivity and Activity Impairment General Health (WPAI-GH) Questionnaire. There are five items (Q1 -Q5) and aimed to measure work productivity namely absenteeism and presenteeism. Absenteeism is defined as the percentage of time miss from work because of LBP and is calculated by the formula Q2/(Q2 + Q4) × 100%. Presenteeism is measured by the degree LBP which affect productivity while working during the past month on a rating scale ranging from 0 " LBP had no effect on my working" to 10 "LBP completely prevented the me from working". Presenteeism is calculated by the formula (Q5/10) × 100%. Outcomes absenteeism and presenteeism are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.

CONTACTS AND LOCATIONS:
Overall Officials: Eva N Zamri, PhD, Principal Investigator — Universiti Sains Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol together its supplement material will be shared with other researchers
Supporting Information: Study Protocol
Time Frame: tentatively May 2024 after publication
Access Criteria: Study Protocol and Supplement Material (Module for Mindfulness for All intervention) will be shared after publication. If other researchers have no access to retrieve the documents, they can request via Principal Investigator's email: evazamri@usm.my